CLINICAL TRIAL: NCT05058534
Title: Impact of a New Multiperfusion Neonatal System on Health and Cost of Care in Neonates
Brief Title: Multiperfusion Neonatal System
Acronym: EDELWEISS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2021_004
Record Dates: First submitted 2021-09-14; First posted 2021-09-27 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Very preterm infants born between November 30, 2018 and November 30, 2019: Infants born between November 30, 2018 - November 30, 2019, before implementation of the new multiperfusion neonatal system
- Very preterm infants born between December 1st, 2019 and December 31st, 2022: Infants born between January 1rst, 2019 - December 31st, 2022, after implementation of the new multiperfusion neonatal system
  Interventions: Device: Multiline Neo®

INTERVENTIONS:
Device: Multiline Neo® — Multiperfusion neonatal system
  Groups: Very preterm infants born between December 1st, 2019 and December 31st, 2022

SUMMARY:
Infusion and parenteral nutrition play an important role in the management of neonatal intensive care patients. Administration of drugs and parenteral nutrition solutions to the patient is performed via different systems including a catheter and a perfusion system. In critically ill, high risk neonates, use of these systems is associated with complications such as infections, interactions between drugs simultaneously infused on the same route (precipitates, catheter obstruction), less effective treatment due to modified amount of drug administered compared to expected or to compatibility issues between drugs. Sepsis and reduction of treatment efficacy can have an impact on survival or subsequent neurodevelopment. Late onset sepsis is one of the most frequent complications in very premature infants born before 33 weeks gestational age and most of those infections occur in infants requiring a perfusion system and an intravenous catheter.

In this context, a new multiperfusion device was developed (Multiline Néo®, Doran, France) to remove access to the infusion system from the incubator where high temperature and humidity favour bacterial growth. But also to allow the administration of several drug solutions simultaneously avoiding contact between drugs.

Our hypothesis is that the new perfusion system helps to reduce the risk of infections, without increase in costs.

ELIGIBILITY:
Inclusion Criteria:

* Born between November 30, 2018 and December 31, 2022,
* Gestational age below 33 weeks

Exclusion Criteria:

* Severe malformation and / or disease requiring heavy surgical management in the neonatal period
* Admitted at croix rousse hospital after the third day of life

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants born between November 30, 2018 and December 31, 2022, at a gestational age below 33 weeks, and hospitalized in the Neonatal unit of Croix-Rousse hospital
Sampling Method: Non-Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Occurence of infection | through study completion, an average of 60 days
  Number of infections per 1000 catheter days, per patient during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civil de Lyon, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared